CLINICAL TRIAL: NCT03555565
Title: Specified Drug-Use Survey of Alogliptin and Metformin Hydrochloride Combination Tablets "Survey on Long-term Use in Type 2 Diabetes Mellitus Patients With Renal or Hepatic Impairment or Advanced Age"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Alogliptin-Met-5003; JapicCTI-183979 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Results first posted 2020-11-23 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin; Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alogliptin and Metformin hydrochloride: Alogliptin 25 mg and metformin hydrochloride 500 mg, combination tablet, orally, once daily for up to 12 months. Participants received interventions as part of routine medical care.
  Interventions: Drug: Alogliptin and Metformin hydrochloride

INTERVENTIONS:
Drug: Alogliptin and Metformin hydrochloride — Alogliptin and Metformin hydrochloride combination tablets
  Other Names: Inisync combination tablets

SUMMARY:
The purpose of this survey is to evaluate the long-term safety and efficacy of the alogliptin and metformin hydrochloride combination tablet in type 2 diabetes mellitus patients with renal impairment (mild), hepatic impairment (mild or moderate), or advanced age (65 years and more) in the routine clinical setting.

DETAILED DESCRIPTION:
The drug being tested in this survey is called alogliptin and metformin hydrochloride combination tablet. This tablet is being tested to treat people who have type 2 diabetes mellitus with renal impairment (mild), hepatic impairment (mild or moderate), or advanced age (65 years and more).

This survey is an observational (non-interventional) study and will look at the long-term safety and efficacy of the alogliptin and metformin hydrochloride combination tablet in the routine clinical setting. The planned number of observed patients will be approximately 600.

This multi-center observational trial will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Participants should meet one or more of the following:

  1. Have renal impairment (mild)
  2. Have hepatic impairment (mild or moderate)
  3. Elderly (aged 65 years or more)

Exclusion Criteria:

* Participants with any contraindication for study drug.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus for whom combination therapy with alogliptin and metformin hydrochloride is appropriate in the opinion of a physician as the routine medical care.
Sampling Method: Probability Sample
Enrollment: 1026 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 115 investigative sites in Japan, from 28 February 2017 to 31 October 2019.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus with renal or hepatic impairment or advanced age were enrolled. Participants received alogliptin and metformin hydrochloride combination tablets as part of a routine medical care.
Period: Overall Study
Arm/Group | Alogliptin and Metformin Hydrochloride
Started | 1026
Completed | 1011
Not Completed | 15
Not completed — Case Report Forms Uncollected | 2
Not completed — Protocol Deviation | 13

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Alogliptin and Metformin Hydrochloride
Number analyzed (Participants) | 1011
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 402
  Male | 609
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 1011
Duration of Diagnosis of Type 2 Diabetes Mellitus [Mean (Standard Deviation); unit: Years] — Mean duration between start of study and first time of diagnosis of type 2 diabetes mellitus was reported. Population: The number analyzed is the number of participants with data available for analysis.
  Years
    number analyzed (Participants) | 663
    (all) | 8.64 (7.297)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 692
    (all) | 66.13 (13.640)
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  Kilogram (kg)/meter (m)^2
    number analyzed (Participants) | 640
    (all) | 25.47 (3.996)
Renal Impairment [Count of Participants; unit: Participants]
  Had No Renal Impairment | 638
  Had Renal Impairment | 373
Hepatic Impairment [Count of Participants; unit: Participants]
  Had No Hepatic Impairment | 545
  Had Hepatic Impairment | 466
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 1006
    Inpatient | 5
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — Number of participants who had or did not have a liability or tendency to suffer from hypersensitivity was reported.
  Participants
    Had No Predisposition to Hypersensitivity | 826
    Had Predisposition to Hypersensitivity | 82
    Unknown | 103
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Medical Complications | 56
    Had Medical Complications | 955
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had No Medical History | 629
    Had Medical History | 267
    Unknown | 115
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 417
  Current Smoker | 156
  Ex-Smoker | 216
  Unknown | 222
Drinking Habits [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported.
  Participants
    Yes | 246
    No | 570
    Unknown | 195
Employment Status [Count of Participants; unit: Participants]
  Not Employed | 495
  Employed | 390
  Unknown | 126
Hemoglobin A1c (HbA1c) Level [Mean (Standard Deviation); unit: Percent] — Population: The number analyzed is the number of participants with data available for analysis.
  Percent
    number analyzed (Participants) | 912
    (all) | 7.336 (1.0710)
Alogliptin-Equivalent Dose per Day Given Immediate Before the Study Drug [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 576
    < 25 milligrams (mg) | 14
    25 mg | 561
    > 25 mg | 1
Metformin-Equivalent Dose per Day Given Immediately Before the Study Drug [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 730
    < 500 mg | 36
    500 mg | 505
    > 500 mg | 189
Combination of Drugs for Type 2 Diabetes Mellitus Other than Alogliptin or Metformin [Count of Participants; unit: Participants]
  Not Combined | 401
  Combined | 610
Status of Treatment Compliance to Alogliptin Medication Within 3 Months prior to the Study Drug [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 558
    ≥ 90% | 487
    ≥ 70% and < 90% | 46
    ≥ 50% and < 70% | 8
    < 50% | 17
Status of Treatment Compliance to Metformin Medication Within 3 Months prior to the Study Drug [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 717
    ≥ 90% | 618
    ≥ 70% and < 90% | 67
    ≥ 50% and < 70% | 17
    < 50% | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had One or More Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: Up to 12 months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Number; unit: Percentage of Participants
Arm/Group | Alogliptin and Metformin Hydrochloride
Number analyzed (Participants) | 1011
Percentage of Participants | 5.93

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at final assessment point (up to Month 12) relative to baseline.
Time Frame: Baseline, up to final assessment point (up to Month 12)
Population: Efficacy assessment population, The efficacy assessment population was defined as participants who completed the survey and had efficacy data at baseline and post-baseline time points available.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Alogliptin and Metformin Hydrochloride
Number analyzed (Participants) | 897
Percent | -0.259 (0.9633)

3. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: The change in the value of fasting blood glucose collected at final assessment point (up to Month 12) relative to baseline.
Time Frame: Baseline, up to final assessment point (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Alogliptin and Metformin Hydrochloride
Number analyzed (Participants) | 468
milligram/deciliter (mg/dL) | -12.08 (46.784)

4. Secondary Outcome: Change From Baseline in Fasting Insulin Level
Description: The change in the value of fasting insulin collected at final assessment point (up to Month 12) relative to baseline.
Time Frame: Baseline, up to final assessment point (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microunit/milliliter (mcrU/mL)
Arm/Group | Alogliptin and Metformin Hydrochloride
Number analyzed (Participants) | 34
microunit/milliliter (mcrU/mL) | 1.21 (13.852)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Alogliptin and Metformin Hydrochloride
All-Cause Mortality (participants affected / at risk) | 1/1011
Serious Adverse Events (participants affected / at risk) | 4/1011
Other Adverse Events (participants affected / at risk) | 13/1011
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin and Metformin Hydrochloride (N=1011)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Atrial fibrillation (Cardiac disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin and Metformin Hydrochloride (N=1011)
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Bundle branch block right (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Chronic gastritis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Malaise (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT03555565/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT03555565/SAP_001.pdf